CLINICAL TRIAL: NCT06764667
Title: Comparison of Spinal Anesthesia Adjuvant and Quadratus Lumborum Block on the Opioid Requirement and Perioperative Pain of Laparoscopic Kidney Transplant Donor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Prof. Dr. dr. Dita Aditianingsih, Sp.An-TI., Subsp.T.I.(K)., Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes048
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Laparoscopic Donor Nephrectomy; Perioperative Pain Management
Keywords: Quadratus lumborum block; Spinal anesthesia adjuvant; Laparoscopic donor nephrectomy; Perioperative pain management
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadratus lumborum block (Active Comparator): Patients in this arm will receive quadratus lumborum block with 20-30 ml of 0.25% Bupivacaine after induction of anesthesia and after operation.
  Interventions: Procedure: Quadratus Lumborum Block (QLB); Procedure: General Anesthesia
- Spinal anesthesia adjuvant (Experimental): Patients in this arm will receive 10 mg 0.5% hyperbaric Bupivacaine, 100 mcg Morphine, 100 mcg Sulfas Atropine, and 0.9% normal saline to total volume of 4 ml before induction of anesthesia.
  Interventions: Procedure: Spinal anesthesia adjuvant; Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Spinal anesthesia adjuvant — Patients in this arm will receive 10 mg 0.5% hyperbaric Bupivacaine, 100 mcg Morphine, 100 mcg Sulfas Atropine, and 0.9% normal saline to total volume of 4 ml before induction of anesthesia.
  Arms: Spinal anesthesia adjuvant
Procedure: Quadratus Lumborum Block (QLB) — Patients in this arm will receive quadratus lumborum block with 20-30 ml of 0.25% Bupivacaine after induction of anesthesia and after operation.
  Arms: Quadratus lumborum block
Procedure: General Anesthesia — The subject will undergo preoxygenation with 100% oxygen for 3 minutes. Following preoxygenation, anesthesia induction will be performed using lidocaine at a dose of 1.5 mg/kg, fentanyl at 1.5 mcg/kg, and propofol at 2.0 mg/kg. Once the subject is adequately sedated, baseline neuromuscular monitoring using the train-of-four (TOF) technique will be conducted, followed by the administration of rocuronium at a dose of 0.8 mg/kg. Endotracheal intubation will be performed using direct laryngoscopy once the TOF value reaches 0, utilizing an appropriately sized endotracheal tube (ETT). Ten milligrams of intravenous dexamethasone is administered after induction.

SUMMARY:
This study aims to compare the effectiveness of spinal anesthesia adjuvant and quadratus lumborum block on the opioid requirement and perioperative pain on patients undergoing laparoscopic kidney transplant donor.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years undergoing laparoscopic donor nephrectomy
* Patients with BMI ≤ 35 kg/m2
* Patients with American Society of Anesthesiology (ASA) physical status 1-2
* Patients who are willing to participate in this study

Exclusion Criteria:

* Cardiovascular disease (uncontrolled stage 2 hypertension, heart failure, arrhytmia)
* Recent onset cerebrovascular diseasae of < 3 months
* Infection on spinal site
* Coagulopathy
* Elevated intracranial pressure
* Severe renal or liver dysfunction
* Valvular heart disease or atrioventricular block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Hour 2, 6, 12, and 24
  Postoperative pain measured with Numerical Rating Scale (NRS) during rest and movement.
Opioid requirement | Hour 2, 6, 12, and 24
  Morphine requirement on Patient-Controlled Analgesia (PCA).

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP dr. Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia